CLINICAL TRIAL: NCT04676347
Title: Evaluation and Improvement of the Health-care Quality in Semi-intensive Care Units
Brief Title: Health-care Quality in Semi-intensive Care Units
Status: Recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: IRFMN_7998
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Semi-intensive Care Unit; Evaluation; Quality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Eligible population: All patients admitted in the semi-intensive care units attending the study. Be basing on the average number of patients yearly treated in those units, we expect to have at least 39000 patients during the 5 years of the study.

SUMMARY:
The main aim of this study is to realize a system of continuous evaluation of healthcare quality in semi-intensive care units.

DETAILED DESCRIPTION:
Collecting data of semi-intensive care units' patients and structural data of hospitals, healthcare quality's indicators will be realized. Starting from those indicators of insuccess, specific for different kinds of patients, it will be possibile to evaluate the general level of care in each singular semi-intensive care unit. The study will least for 5 years, but at the end of every year it will be realized a report of analysis to see the results of each unit.

ELIGIBILITY:
Inclusion Criteria:

* all patients hospitalised in a semi-intensive care unit

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients hospitalised in a semi-intensive care unit attending the study, during a 5 years period of time (from 1st january 2021, to 31st december 2025)
Sampling Method: Non-Probability Sample
Enrollment: 39000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Outcome for stationary patients with high risk of variability | jan 2021 - dec 2025
  hospitalization in semi-intensive care unit more than 2 days or transfer to intensive care unit
Outcome for low gravity patients, with a low organ's damage | jan 2021 - dec 2025
  deterioration of the physiopathologic index
Outcome for semi-intensive patients | jan 2021 - dec 2025
  transfer to intensive care unit or hospital mortality
Outcome for high risk patients | jan 2021 - dec 2025
  transfer to intensive care unit or hospital mortality

CONTACTS AND LOCATIONS:
Locations (25):
- Italy (25):
  - Istituto di Ricerche Farmacologiche Mario Negri IRCCS, Milan, Milan
  - ASO SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - Ospedale Umberto Parini, Aosta
  - Ospedale San Bassiano, Bassano del Grappa
  - Ospedale Maggiore, Bologna
  - AOU Policlinico S. Marco, Catania
  - AOU Policlinico San Marco, Catania
  - Ospedale Bufalini, Cesena
  - Ospedale Santa Maria Annunziata, Florence
  - Ospedale Morgagni-Pierantoni, Forlì
  - Ospedale Palmanova-Latisana, Latisana
  - Ospedali Riuniti, Livorno
  - ASST Lodi, Lodi
  - Ospedale Santa Maria delle Grazie, Napoli
  - AOU San Luigi Gonzaga, Orbassano
  - Ospedale Guglielmo da Saliceto, Piacenza
  - Ospedale E.Agnelli, Pinerolo
  - AOU Pisana, Pisa
  - Ospedale Santa Maria delle Croci, Ravenna
  - Ospedale Sant'Eugenio, Roma
  - AOU di Sassari, Sassari
  - Ospedale Giovanni Bosco, Torino
  - Ospedale Ca' Foncello, Treviso
  - Santa Maria della Misericordia, Udine
  - Ospedale Michele e Pietro Ferrero, Verduno

IPD SHARING:
Plan to Share IPD: Undecided
Protecting the privacy policy, all the data that underlie results in a publication will be shared. The scientific commettee of the study has to decide the criteria and the best way to share them